CLINICAL TRIAL: NCT01991756
Title: ELEVATE International: Kissing Endografts for Peripheral AAA Exclusion
Brief Title: Safety and Performance of Altura Endograft in Abdominal Aortic Aneurysm (AAA) Endovascular Repair
Acronym: ELEVATE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Altura Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALTURA-ELE-1
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Abdominal Aortic Aneurysms; AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AAA: Subjects with a documented untreated, unruptured, infrarenal abdominal aorto-iliac aneurysm will be treated with the Altura Endograft System.
  Interventions: Device: Altura Endograft System

INTERVENTIONS:
Device: Altura Endograft System — Subjects with a documented untreated, unruptured, infrarenal abdominal aorto-iliac aneurysm.

SUMMARY:
The primary objective of the study is to evaluate the acute safety of deploying and implanting the Altura Endograft in the treatment of AAA in subjects who are candidates for endovascular repair.

Secondary objectives are to evaluate the acute and longer-term safety and performance of the Altura Endograft through 5 years.

DETAILED DESCRIPTION:
The primary safety endpoint of the study is freedom from Major Adverse Events (MAE), a composite endpoint consisting of death, stroke, paraplegia, myocardial infarction, respiratory failure, renal failure, bowel ischemia and blood loss ≥ 1000 mL.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Understands and has signed an Informed Consent
* Candidate for endovascular or open surgical repair of an infrarenal aortic or aorto-iliac aneurysm
* Abdominal aneurysm > 45 mm or aneurysm growth of > 10 mm/year
* Abdominal aneurysm neck angulation ≤ 60 degrees
* Infrarenal non-aneurysmal neck 15 mm
* Infrarenal non-aneurysmal neck diameter between 18 and 28 mm, inclusive
* Iliac artery landing zone 15 mm in length
* Iliac artery landing zone diameter between 8 and 18 mm, inclusive
* Patent iliac and femoral arteries, access vessels, size and morphology, to allow endovascular access of a minimum 14 Fr introducer sheath and catheter
* Ability to preserve at least one hypogastric artery
* Life expectancy > one year
* American Society of Anesthesiology (ASA) grade 1 through 3, inclusive
* Able and willing to comply with follow-up visits at 30 days, 6 and 12 months and annually through 5 years

Exclusion Criteria:

* Pregnant or nursing
* An acutely ruptured, leaking or emergent aneurysm
* An aortic dissection (Type A or B)
* A mycotic, infected or inflammatory aneurysm
* A thoracic, suprarenal or juxtarenal aneurysm
* Previous surgical or endovascular aneurysm repair for abdominal aortic aneurysm or an aorto-iliac aneurysm
* Severe iliac artery tortuosity
* Thrombus, calcification and/or plaque that may complicate sealing
* Evidence or history of intracranial bleeding or aneurysm, myocardial infarction or stroke within the past 3 months
* Current angina or other active cardiac condition such as congestive heart failure, untreated or worsening atrial arrhythmia, ventricular arrhythmia or valvular disease
* Had or plans to have an unrelated major surgical or interventional procedure within 1 month before or after implantation of the study device
* Significant (>80%) diameter renal artery stenosis which could not be readily treated
* Known sensitivity or allergy to nitinol or polyester
* Known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment
* Contraindication to antiplatelet, anticoagulant or thrombolytic therapy;
* Coagulopathy or uncontrolled bleeding disorder
* History of heparin-induced thrombocytopenia (HIT)
* Clinically and morbidly obese such that the required imaging would be prevented
* Connective tissue disease (e.g., Marfan's or Ehlers-Danlos syndromes)
* Currently on dialysis or has compromised renal function as reflected by a serum creatinine >2.0 mg/dL
* Compromised hepatic function
* Active infection at the time of the index procedure
* End-stage chronic obstructive pulmonary disorder (COPD)
* Religious, cultural or other objections to the receipt of blood or blood products
* Participating in another research study involving an investigational device or drug which may potentially affect study results
* Other medical, social or psychological problems that, in the opinion of the Investigator, preclude them from receiving this treatment and the procedures and evaluations pre- and post-treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with infrarenal abdominal aortic aneurysm (AAA) disease with suitable aneurysm morphology for endovascular repair.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 30 days
  Freedom from Major Adverse Events (MAE), a composite endpoint consisting of:
  * Death
  * Stroke
  * Paraplegia
  * Myocardial infarction
  * Respiratory failure
  * Renal failure
  * Bowel ischemia
  * Blood loss ≥ 1000 mL

SECONDARY OUTCOMES:
Secondary Safety Endpoint | 30 days, 6 and 12 months and annually through 5 years
  * Major Adverse Events (MAE)
  * Aneurysm-related death
  * Type I and III endoleaks
  * AAA rupture
  * Re-intervention to correct Type I or Type III endoleaks, migration, occlusion, narrowing, stenosis, kinking or fracture

OTHER OUTCOMES:
Secondary Performance Endpoint | Procedurally, 30 days, 6 and 12 months and annually through 5 years
  * Acute Technical Success
  * Longer-term Technical Success, defined as subjects having Acute Technical Success and no evidence of
    * Migration (greater than or equal to 10 mm)
    * Occlusion
  * Clinical Success, defined as subjects having Acute Technical Success and no evidence of
    * Type I or Type III endoleaks
    * AAA rupture
    * Re-intervention (surgical or endovascular) to correct Type I or Type III endoleaks, migration, occlusion, narrowing, stenosis, kinking or fracture.
  * Change in aneurysm sac size diameter
    * Absolute change (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, PhD, Principal Investigator — Park-Krenkenhaus Leipzig
Locations (4):
- Germany (4):
  - Uniklink, Freiburg im Breisgau
  - University Heart Center, Hamburg-Eppendorf
  - Park-Krankenhaus Leipzig, Leipzig
  - Sankt Bonifatius Hospital, Lingen